CLINICAL TRIAL: NCT05221580
Title: A Prospective Non-interventional Single-arm Study Investigating Clinical Parameters Associated With the Use of Ryzodeg® (Insulin Degludec/Insulin Aspart) in a Real-world Adult Population With Type 2 Diabetes in China
Brief Title: China Research of IDEgAsp Treatment in Real-world Clinical practicE (CREATE)
Acronym: CREATE
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN5401-4623; U1111-1238-6960 (Other: World Health Organization (WHO))
Record Dates: First submitted 2022-01-12; First posted 2022-02-03 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — insulin degludec, insulin aspart drug combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Real-world adult population of Chinese patients with T2DM: Ryzodec as per local clinical practise
  Interventions: Drug: Ryzodeg®

INTERVENTIONS:
Drug: Ryzodeg® — Patients will be treated with commercially available Ryzodeg® in a prefilled device (FlexTouch®) or in a penfill according to the label and routine clinical practice at the discretion of the treating physician

SUMMARY:
The purpose of this study is to collect information on how Ryzodeg® works in real-world patients.

Participants will get Ryzodeg® as prescribed to by their doctor. The study will last for about 5-8 months. Participants will be asked questions about their health and their diabetes treatment as part of their normal doctor's appointment

ELIGIBILITY:
Inclusion Criteria:

1. Signed consent obtained before any study-related activities (study-related activities are any procedure related to recording of data according to the protocol).
2. The decision to initiate treatment with commercially available Ryzodeg® has been made by the patient/Legally Acceptable Representative (LAR) and the treating physician based on the approved Ryzodeg® label in China and independently from the decision to include the patient in this study.
3. Male or female, age above or equal to 18 years at the time of signing informed consent.
4. Diagnosed with T2DM and treated with any anti-hyperglycaemic medication(s) other than Ryzodeg® for at least 20 weeks prior to Treatment Initiation Visit (Visit 1).
5. Available and documented Glycosylated haemoglobin (HbA1c) value below or equal to 12 weeks prior to Informed Consent and Treatment Initiation Visit (Visit 1).

Exclusion Criteria:

1. Previous participation in this study. Participation is defined as having given informed consent in this study.
2. Treatment with any investigational drug within 30 days prior to enrolment into the study.
3. Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation.
4. Known or suspected hypersensitivity to the active substance or to any of the excipients as specified in the approved Ryzodeg® label in China.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Real-world adult population with type 2 diabetes in China.
Sampling Method: Non-Probability Sample
Enrollment: 887 (Actual)
Dates: Start 2022-03-18 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Change in Glycosylated Haemoglobin (HbA1c) | From baseline (week 0) to end of study (week 20 to 32)
  Percentage point

SECONDARY OUTCOMES:
HbA1c less than 7 percent (Yes/No) | At the end of study (week 20 to 32)
  Percentage of patients
HbA1c less than 7 percent without any hypoglycaemic episodes during 4 weeks prior to end of study (Yes/No) | At the end of study (week 20 to 32) Hypoglycaemic episodes occurring within 4 weeks prior to end of study (week 20 to 32).
  Percentage of patients
Change in Fasting Plasma Glucose (FPG) | From baseline (week 0) to end of study (week 20 to 32)
  mmol/L
Change in insulin dose (total, basal, prandial) | From baseline (week 0) to end of study (week 20 to 32)
  units/day
Change in body weight | From baseline (week 0) to end of study (week 20 to 32)
  Kg
Patient preference compared to previous treatment | At baseline and end of study (week 20 to 32)
  Percentage of patients who prefer to continue treatment with Ryzodeg® over previous treatment. Assessed by questionnaire
Treatment satisfaction questionnaire (Diabetes Treatment Satisfaction Questionnaire (DTSQ)) | At baseline and end of study (week 20 to 32)
  Score based on items 1, 4, 5, 6, 7 and 8. Range 0-36, where higher score means greater satisfaction (better outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (50):
- China (50):
  - NIS-The Second People's Hospital of Hefei, Hefei, Anhui
  - NIS-Beijing Hospital, Beijing, Beijing Municipality
  - NIS-Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - NIS-People's Hospital of Chongqing Banan District, Chongqing, Chongqing Municipality
  - NIS-Gansu Provincial People's Hospital, Lanzhou, Gansu
  - NIS-The people's hospital of JiangMen, Jiangmen, Guangdong
  - NIS-2nd Affiliated Hospital of Shantou University Medical, Shantou, Guangdong
  - NIS-Shenzhen Longgang District People's Hospital, Shenzhen, Guangdong
  - NIS-Yangjiang People's Hospital, Yangjiang, Guangdong
  - NIS-The First People's Hospital of Yulin City, Yulin, Guangxi
  - NIS-Hainan Provincial Hospital of TCM, Haikou, Hainan
  - NIS-Cangzhou Hosp of Integrated Traditional Chinese Medicine, Cangzhou, Hebei
  - NIS-The First Hospital of Handan, Handan, Hebei
  - NIS-The First Hospital of Qinhuangdao, Qinhuangdao, Hebei
  - NIS-Heilongjiang Provincial Hospital, Harbin, Heilongjiang
  - NIS-Zhengzhou University - The Second Affiliated Hospital, Zhengzhou, Henan
  - NIS-Shiyan City People's Hospital, Shiyan, Hubei
  - NIS-Puai Hospital of Wuhan, Wuhan, Hubei
  - NIS-The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - NIS-The Sceond Hospital of Chifeng, Chifeng, Inner Mongolia
  - NIS-Inner Mongolia University for Nationalities - Affiliated, Tongliao, Inner Mongolia
  - NIS-Changshu Second People's Hospital, Changshu, Jiangsu
  - NIS-Huai'an First People's Hospital, Huai'an, Jiangsu
  - NIS-Nanjing Jiangning Hospital, Nanjing, Jiangsu
  - NIS-Jiangsu Province Officeial Hospital, Nanjing, Jiangsu
  - NIS-Nantong University - Affiliated Hospital, Nantong, Jiangsu
  - NIS-Yixing City People's Hospital, Yixing, Jiangsu
  - NIS-Affiliated Hospital of Jilin Medical College, Jilin, Jilin
  - NIS-Songyuan Jilin Oilfield Hospital, Songyuan, Jilin
  - NIS-The Third People's Hospital of Dalian, Dalian, Liaoning
  - NIS-Huludao Central Hospital, Huludao, Liaoning
  - NIS-Third Affiliated Hospital of Jinzhou Medical University, Jinzhou, Liaoning
  - NIS-The Fourth Hospital of China Medical University, Shenyang, Liaoning
  - NIS-The People's Hospital of Ningxia Hui Autonomous Region, Yinchuan, Ningxia
  - NIS- Qinghai Red Cross Hospital, Xining, Qinghai
  - NIS-Hanzhong Central Hospital, Hanzhong, Shaanxi
  - NIS-Shanxi Bethune Hospital, Taiyuan, Shaanxi
  - NIS-Xi'an No.3 Hospital, Xi'an, Shaanxi
  - NIS-Weifang Medical University - Affiliated Hospital, Weifang, Shandong
  - NIS-Binzhou Medical University-Yantai Affiliated Hospital, Yantai, Shandong
  - NIS-Central hospital of zibo, Zhibo, Shandong
  - NIS-Shanghai Shidong Hospital, Shanghai, Shanghai Municipality
  - NIS-Shanghai Shuguang Hospital, Shanghai, Shanghai Municipality
  - NIS-Affiliated Hospital of North Sichuan Medical College, Nanchong, Sichuan
  - NIS-Metabolic Diseases Hosp&Tianjin Institute of Endocrinolo, Tianjin, Tianjin Municipality
  - NIS-Tianjin First Center Hospital, Tianjin, Tianjin Municipality
  - NIS-De Hong Zhou People's Hospital, Mang City, Yunnan
  - NIS-The First People's Hospital of Qujing, Qujing, Yunnan
  - NIS-Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang
  - NIS-Shaoxing Central Hospital, Shaoxing, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com